CLINICAL TRIAL: NCT05319275
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of Acetyllevocarnitine Hydrochloride Tablets in Chinese Patients With Paresthesias Caused by Diabetic Peripheral Neuropathy
Brief Title: Study of Acetyllevocarnitine Hydrochloride Tablets in Chinese Patients With Paresthesias Caused by DPN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Heisco19-301
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Peripheral Neuropathy (DPN); Paresthesia
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetyllevocarnitine Hydrochloride Tablets (Experimental)
  Interventions: Drug: Acetyllevocarnitine Hydrochloride Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetyllevocarnitine Hydrochloride Tablets — 500 mg (2×250 mg/tablet) after meal, 3 times per day
  Arms: Acetyllevocarnitine Hydrochloride Tablets
Drug: Placebo — 500 mg (2×250 mg/tablet) after meal, 3 times per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Acetyllevocarnitine Hydrochloride Tablets compared with placebo after 24 weeks, in chinese patients with paresthesia caused by Diabetic Peripheral Neuropathy (DPN).

DETAILED DESCRIPTION:
This 24-week, multicentre, randomised, double-blind, placebo-controlled phase III study is to assess the efficacy and safety of Acetyllevocarnitine Hydrochloride Tablets in Chinese patients with paresthesia caused by DPN.The trial included a 2-week screening period, a 1-week placebo run-in period, a 24-week randomized treatment period, and a 2-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 years, Male and female patients;
* Type 1 or 2 diabetes mellitus on hypoglycemic therapy for 3 months or more, and clinical diagnosis of DPN;
* HbA1c < 9.0%;
* Toronto Clinical Neuropathy Score ≥ 6 at screening and baseline.

Exclusion Criteria:

* Peripheral neuropathy caused by other diseases;
* History of acute complications of diabetes within the past 6 months, such as diabetic ketoacidosis, diabetic hyperosmolar hyperglycemia syndrome or lactic acidosis, etc.;
* Severe peripheral arterial disease; severe cardiopulmonary disease; or have a history of myocardial infarction, cerebrovascular accident or transient ischemic attack within 6 months before enrollment; or uncontrolled asthma or shortness of breath 2 months before enrollment; World Health Organization (WHO) cardiac function class III-IV; systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg at screening;
* Any infection at the screening visit that is not suitable for study participation;
* Aspartate Transaminase (AST) or Alanine Transaminase (ALT) or total bilirubin or creatinine > 2 times Upper Limit of Normal (ULN);
* Known allergy to L-carnitine ingredients;
* Severe systemic or psychiatric illness, history of epilepsy;
* History of malignancy or antitumor therapy;
* Severe bleeding disorder;
* Clinically significant abnormalities in thyroid function tests;
* Triglyceride >5.6 mmol/L;
* Change of 2 points or more in the same item in mTCNS;
* Nursing or pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
mTCNS total score change from baseline at week 24 | Baseline and week 24
  Changes in Modified Toronto Clinical Neuropathy Score (mTCNS) total score from baseline at Week 24. Maximum mTCNS is 33, minimum is 0. And higher points mean more serious condition. However, more points drop from baseline mean a better outcome.

SECONDARY OUTCOMES:
mTCNS total score change from baseline at week 12 | Baseline and week 12
  Changes in Modified Toronto Clinical Neuropathy Score (mTCNS) total score from baseline at Week 12. Maximum mTCNS is 33, minimum is 0. And higher points mean more serious condition. However, more points drop from baseline mean a better outcome.
Changes in each item score of mTCNS from baseline at week 12 and week 24 | Baseline, Weeks 12 and 24
  The mTCNS contains the 11 items that assess symptoms and signs, and each item maximum is 3 points, minimum is 0. And higher points mean more serious condition. However, more points drop from baseline mean a better outcome.
TCNS total score change from baseline at week 12 and week 24 | Baseline, Weeks 12 and 24
  Changes in Toronto Clinical Neuropathy Score (TCNS) total score from baseline at Week 12 and Week 24. Maximum TCNS is 19, minimum is 0. And higher points mean more serious condition. However, more points drop from baseline mean a better outcome.
Numeric Rating Scale (NRS) score change from baseline at week 24 | Baseline and week 24
  Changes in Numeric Rating Scale (NRS) score from baseline at Week 24. Maximum NRS is 10, minimum is 0. And higher points mean more serious condition. However, more points drop from baseline mean a better outcome.
Changes in Nerve Conduction Velocity (NCV) from baseline at week 24 | Baseline and week 24
Changes in Nerve Conduction Amplitude from baseline at week 24 | Baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Guo, Study Chair — Beijing Hospital
Locations (34):
- China (34):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan Third People's Hospital, Sanya, Hainan
  - Handan Central Hospital, Handan, Hebei
  - Hebei Petro China Center Hospital, Langfang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Kaifeng Traditional Chinese Medicine Hospital, Kaifeng, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Medical Group of Zhengzhou First People's Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiujiang Traditional Chinese Medicine Hospital, Jiujiang, Jiangxi
  - The Fourth Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Yichun People's Hospital, Yichun, Jiangxi
  - Affiliated Hospital of Yanbian University, Yanbian, Jilin
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Chongqing People's Hospital, Chongqing
  - Yongchuan Hospital of Chongqing Medical University, Chongqing
  - Tianjin First Central Hospital, Tianjin